CLINICAL TRIAL: NCT04252755
Title: Enhancing Brain Processing Via Neurofeedback in Addictive Disorders: A Pilot Study
Brief Title: Enhancing Brain Processing Via Neurofeedback in Addictive Disorders
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped prior to initiation due to COVID-19 complications
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HIREB#8178
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Alcohol Drinking
Keywords: Electroencephalography (EEG); Neurofeedback; Alcohol Use; Cognition
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: This study will utilize a pre-post within-subjects design. All participants will undergo a baseline (pre) session, then be scheduled for 8 sessions of neurofeedback, and finish with another session (post) after completion of all neurofeedback sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EEG Neurofeedback (Other): Within-subjects sessions of EEG neurofeedback
  Interventions: Behavioral: EEG Neurofeedback

INTERVENTIONS:
Behavioral: EEG Neurofeedback — Participants will undergo a baseline (pre) session, then be scheduled for 8 sessions of NFB, and finish with another session (post) after completion of all NFB sessions.

SUMMARY:
The purpose of this study is to investigate the effects of neurofeedback training on measures of cognitive control and alcohol motivation among young adults who drink alcohol on a regular basis. Neurofeedback is a cognitive training technique that uses portable electroencephalography (EEG) technology to adjust brain activity through immediate sensory feedback. This study is using a type of EEG device called a MuseTM headset that monitors ongoing brain activity and synchronizes this information with a mindfulness training app on a mobile device. This study is a pilot study to examine the feasibility and effects of neurofeedback training in a sample of young adults. Future studies may use similar protocols with people who have substance use disorders or other mental health disorders.

DETAILED DESCRIPTION:
The NFB studies conducted to date have utilized a wide range of methodologies and NFB training protocols. The outcome measures of NFB efficacy have also varied widely. As mentioned above, the studies also used expensive, non-portable equipment which may limit the application of NFB in treatment settings. This study seeks to address these limitations by using a commercially-available neurotechnology, the Muse™ headband by InteraXon (Toronto, ON, Canada) and using their standard NFB protocol built into the device application. This will maximize the standardization and portability of the NFB as essentially an "out of the box" intervention. The outcome measures will also capture multiple relevant domains, including clinical outcomes (e.g., drinking motivation) and neurocognitive performance (e.g., cognitive control / response inhibition).

The purpose of this study is to investigate the effects of NFB training on measures of cognitive control and alcohol motivation among young adults who engage in heavy episodic drinking (defined as exceeding 4+/5+ drinks per occasion for men/women).

The study will examine whether NFB reduces motivation/attention and craving for alcohol and attentional bias to alcohol-related cues. The primary outcome will be assessed by changes in the alcohol purchase task and approach/avoidance task, which participants will complete pre- and post-NFB training.

A secondary outcome is to determine whether NFB results in transfer of heightened fronto-cortical activity to improvements on general executive functioning following 8 sessions of NFB training. The secondary outcome will be assessed via changes in neurocognitive tasks assessing behavioural inhibition, risky decision making, and executive functioning, all of which will be administered pre- and post-NFB training.

ELIGIBILITY:
Inclusion Criteria:

* Current undergraduate student, can be registered in the SONA research participant pool
* 18 years or older
* At least one self-reported heavy drinking episode in the last two weeks (e.g., consumption of 5/4+ alcoholic drinks in a single drinking episode for men/women).

Exclusion Criteria:

* History of stroke, seizures, or traumatic brain injury
* Any history of severe psychiatric disorders, including schizophrenia-spectrum, bipolar disorder, Post-traumatic stress disorder.
* Presence of skin conditions/headwear that cannot be removed on the forehead/scalp that could interfere with EEG signal (e.g., open cuts, eczema, heavy acne, or psoriasis)
* Greater than weekly use of cannabis or greater than monthly use of other illicit drugs (e.g. cocaine, methamphetamine, opioids, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Alcohol motivation | 14 days
  Alcohol demand will be assessed via a hypothetical purchase task measuring self-reported consumption of alcohol across a range of prices. Primary dependent measure of this task is the amount of alcohol purchased and money spent.
Alcohol approach/avoidance bias | 14 days
  Approach-avoidance bias will be assessed via an implicit approach/avoidance task involving pushing or pulling images closer/farther away using a joystick. Primary dependent measure from this task is latency of response to alcohol vs. neutral images for the approach and avoidance conditions.
Alcohol craving | 14 days
  Subjective alcohol craving will be assessed via a visual analog scale (0-100, with 100 equal to maximum craving)

SECONDARY OUTCOMES:
Behavioural inhibition | 14 days
  Behavioural inhibition will be assessed via computerized task of inhibitory control (go/no-go task) requiring suppression of inappropriate behavioural responses to "no-go" cues. Primary dependent measure is the percentage of correct trials and percentage of inhibitory failures
Risky decision-making | 14 days
  Risky decision making will be assessed via a Balloon Analogue Risk Task involving pumping a hypothetical balloon with an unknown air capacity. Each pump results in greater points earned, but a popped balloon results in loss of all accumulated points. Primary dependent variable from this task is the total number of pumps and number of exploded balloons. Higher values for each variable reflect greater risk taking
Interference control | 14 days
  Interference control will be assessed via the Erikson Flanker Task involving making a behavioural response to a central stimulus (left/right arrow) that is flanked by arrows that either point in same direction (congruent) or opposite direction (incongruent). Primary dependent variable is the percentage of correct trials in congruent vs incongruent conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Amlung, PhD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada